CLINICAL TRIAL: NCT02496234
Title: The Use of Aging Biomarkers to Predict Adverse Outcomes After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Sapere Bio (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: HSDX-1503
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Bypass Graft Surgery; Acute kidney injury; Renal failure; Biomarker
MeSH Terms: conditions — Coronary Artery Disease; Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — White blood cells Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiac surgery associated acute kidney injury (CSA-AKI) has been recognized as the second most common cause of hospital acquired AKI. The development of CSA-AKI is independently associated with an increased risk of in-hospital death. There are currently no biomarkers that could identify patients at higher risk for AKI and current risk predictor scores that are based on clinical and demographic information are inadequate. Therefore, a diagnostic test for predicting AKI risk in this clinical context would assist clinicians to optimize surgical strategy and postoperative care to prevent CSA-AKI occurrence and improve patient outcomes.

The primary purpose of this study is to measure the association between baseline expression of senescence markers in blood using SenesceTest and the occurrence of CSA-AKI post surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all criteria to be eligible for this study:

* Adult patients (>18 yo) undergoing non-emergency cardiac surgery using cardiopulmonary bypass (CABG, combined CABG/valve, or valve surgery).

Exclusion Criteria:

Patients who fulfill any of the following criteria will be excluded:

* Emergency surgery.
* Off-pump coronary bypass grafting.
* Aortic aneurysm repair.
* Congenital heart disease repair.
* Heart transplant or LVAD patient.
* Severe heart failure (LVEF<25%).
* Hemodynamic instability or requiring preoperative vasopressors or IABP.
* Pre-existing end-stage kidney disease (eGFR< 15 mL/min/1.73 m2) or renal transplantation.
* Presence of major active infection (chronic or acute, e.g. sepsis, HIV, pneumonia).
* Chronic liver disease /cirrhosis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects entered into this study will be patients of the Duke University Health System.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Development of stage 1 or higher postoperative AKI as defined by the AKIN classification (stage 1- ≥ 0.5 mg/dL absolute or ≥ 50% relative rise in peak SCr over the baseline) | 48-72 hours

SECONDARY OUTCOMES:
Number of Participants who suffered postoperative stroke | 30 days
Number of Participants who suffered cognitive decline | 30 days
Number of Participants requiring prolonged mechanical ventilation (for longer than 24h) | 30 days
Number of Participants with : cardiac arrest, perioperative myocardial infarction and perioperative ventricular dysfunction. | 30 days
Number of Participants with cardiac arrest | 30 days
Number of Participants with perioperative myocardial infarction | 30 days
Number of Participants with perioperative ventricular dysfunction. | 30 days
Number of Participants with postoperative deep sternal wound infection | 30 days
Number of Participants with postoperative thoracotomy infection | 30 days
Number of Participants with postoperative sepsis. | 30 days
Number of Participants in need for renal replacement therapy | 30 days
Number of Participants who progressed to end stage renal disease. | 30 days
Death | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mihai V Podgoreanu, MD, FASE, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States